CLINICAL TRIAL: NCT02082405
Title: A Phase II Trial of Weekly Bortezomib and Dexamethasone With Oral Metronomic Cyclophosphamide in Elderly Patients With Plasma Cell Myeloma
Brief Title: Bortezomib, Dexamethasone, and Cyclophosphamide in Treating Older Patients With Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3A13; NCI-2014-00250 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 3A13 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cyclophosphamide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bortezomib, cyclophosphamide, dexamethasone) (Experimental): Patients receive bortezomib SC or IV over 3-5 seconds on days 1, 8, and 15; cyclophosphamide PO QD on days 1-21; and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Drug: cyclophosphamide; Drug: dexamethasone; Other: laboratory biomarker analysis; Other: quality-of-life assessment

INTERVENTIONS:
Drug: bortezomib — Given SC or IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: cyclophosphamide — Given PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Other: laboratory biomarker analysis — Optional correlative studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase II trial studies the side effects and how well lower doses of bortezomib, dexamethasone, and cyclophosphamide work in treating older patients with multiple myeloma. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving cyclophosphamide daily may kill more cancer cells. Giving bortezomib, cyclophosphamide, and dexamethasone may be an effective treatment for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR) and toxicity rate of therapy with weekly bortezomib combined with oral metronomic cyclophosphamide and low-dose dexamethasone.

SECONDARY OBJECTIVES:

I. To determine overall survival. II. To describe the association between disease status, treatment response, treatment toxicity, quality of life, functional status, risk for development of frailty, and inflammatory cytokine levels.

OUTLINE:

Patients receive bortezomib subcutaneously (SC) or intravenously (IV) over 3-5 seconds on days 1, 8, and 15; cyclophosphamide orally (PO) once daily (QD) on days 1-21; and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of symptomatic myeloma in accordance with International Myeloma Working group (IMWG) criteria

  * Bone marrow plasmacytosis with > 10% plasma cells or sheets of plasma cells or biopsy proven plasmacytoma
  * Symptomatic disease, i.e., end-organ damage due to multiple myeloma (MM) including at least one of the following: anemia, hypercalcemia, bone disease (lytic bone lesions or pathologic fracture), or renal dysfunction
* Absolute neutrophil count (ANC) >= 1000 cells/mm^3 (without use of growth factors)
* Platelets >= 50,000 cells/mm^3
* Direct bilirubin =< 1.5 X upper limit of normal (ULN); elevated bilirubin is permissible if patient has a known history of elevated bilirubin due to Gilbert's or if elevated bilirubin is due to hemolysis
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 X ULN
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior treatment with > 1 cycle of any plasma cell myeloma (PCM) induction regimen (maximum 6 weeks of prior treatment)

  * Prior radiation therapy is allowed
  * Prior treatment for other cancers is allowed as long as patient meets criteria for adequate hematopoietic and organ function and is not actively on chemotherapy for another cancer
* Grade >= 2 peripheral neuropathy
* Second malignancy currently undergoing chemotherapy or radiotherapy; hormonal therapy for breast or prostate cancer is allowed
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib, cyclophosphamide, dexamethasone or other agents used in this study
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Overall Response rate in accordance with the IMWG Uniform Response criteria | Up to 7 months
  The number of people with any response as defined by the IMWG criteria
Incidence of toxicities according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4 | Up to 7 months

SECONDARY OUTCOMES:
Changes in quality of life as assessed by the Functional Assessment of Cancer Therapy-General | Up to 24 weeks
  Changes in quality of life at baseline to the end of treatment estimated by means with confidence intervals. Quality of life will be assessed using the 34 item general functional assessment of cancer therapy (FACT-G) questionnaire.
Changes in functional status | Up to 24 weeks
  Changes in functional status at baseline to the end of treatment estimated by means with confidence intervals. Functional status will be assessed by scoring the thirteen item Vulnerable Elders Survey (VES-13).
Overall Survival | 24 Weeks
  The number of people alive after 24 weeks on the study
Changes in quality of life as assessed by the Functional Assessment of Cancer Therapy-General | After 6 weeks (2 courses) of treatment
  Average changes in quality of life at baseline estimated by means with confidence intervals.Quality of life will be assessed using the 34 item general functional assessment of cancer therapy (FACT-G) questionnaire.
Changes in functional status | After 6 weeks (2 courses) of treatment
  Changes in functional status at baseline to the second course 2 of therapy estimated by means with confidence intervals. Functional status will be assessed by scoring the thirteen item Vulnerable Elders Survey (VES-13).

CONTACTS AND LOCATIONS:
Overall Officials: Erica Campagnaro, Principal Investigator — Case Comprehensive Cancer Center